CLINICAL TRIAL: NCT06595225
Title: Lifestyle and Nutrition Intervention for Patients Living with HIV Attending an Outpatient Clinic in Dubai, UAE
Brief Title: Nutrition Education Intervention for PLHIV
Acronym: 202372
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Souheir Alia, Clinical dietitian and PhD candidate, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202372
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hiv; Nutritional Deficiency
Keywords: Nutrition education; HIV; PLHIV; Intervention; Knowledge. attitude, practices
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Malnutrition

STUDY DESIGN:
Intervention Model Description: Participants were assigned randomly into either the control or intervention group based on 4 aspects which were: gender, 0 co-morbidities, 1 co-morbidity, 2 or more co-morbidities, whereas the interventional group received nutrition education sessions of various topics related to general nutrition knowledge, with more focus on nutrition related to patients living with HIV (PLHIV) for a 6 months period, were there was one encounter per month and follow up was weekly over a social media platform (Whatsapp)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition Education Sessions Group (Experimental): this group received nutrition education sessions each month for a period of 6 months. Where they were followed up once a week via Whatsapp, reminded of the previous session's message and had their questions answered.
  Interventions: Behavioral: Nutrition education sessions
- Control group (No Intervention): this group did not receive the intervention that the experimental group received

INTERVENTIONS:
Behavioral: Nutrition education sessions — Participants received nutrition education each month, covering topics ranging from general nutrition knowledge, nutrition knowledge related to their diagnosis of living with HIV infection whether during the acute or chronic phase. In addition, specific information was shared about other comorbidities the participant could be living with, finally information was shared on ways to improve mental health and enhance physical activity levels.
  Arms: Nutrition Education Sessions Group

SUMMARY:
The study tested two hypotheses, which are mentioned below:

Hypotheses: The project will test 5 hypotheses related to the various aspects of the study.

H1: implementing a nutrition education intervention will significantly improve the patient's nutritional knowledge, dietary practices, and attitudes (KAP) post-6 months of intervention.

H2: implementing a nutrition education intervention will significantly improve the patients' food intake of immune-boosting foods, physical activity levels, anthropometric measurements, nutrition-related biochemical biomarkers, and mental health status, post the intervention period.

Note: H2 is a complex hypothesis consisting of 5 sub-hypotheses corresponding to the five mentioned measurements (food intake of immune-boosting foods, physical activity levels, anthropometric measurements, nutrition-related biochemical biomarkers, and mental health status). Each of these sub-hypotheses will be statistically tested.

DETAILED DESCRIPTION:
The intervention was guided by the Health Belief model. The topics to be covered and the content of the educational program were designed with input from dietitians working with PLHIV to ensure the relevance for the target participants. Participants randomized into the intervention group received individualized sessions with a registered dietitian once a month for 6 months. During the sessions, the dietitian elaborated on the medical nutrition therapy for each participant which consists of nutritional diagnosis and nutritional counseling services. Topics covered include general nutrition knowledge, MyPlate food groups, immune-boosting foods and nutrients, improving physical activity levels, the nutritional aspects of the existing co-morbidities such as hypertension, diabetes, etc. The intervention provided by the dietitian (primary investigator) which was guided by the Health Belief Model (HBM) which suggests that an individual's beliefs about health threats, perceived benefits of acting, and perceived barriers to acting are key determinants of health-related behaviors. Each session lasted for approximately 30-45 minutes through virtual platforms or in-person, or a combination of both, using several teaching tools such as discussions, demonstrations, educational materials, and educational videos.

The participants were met with online once per month and they were followed up on weekly basis on Whatsapp to reinforce the last session message.

ELIGIBILITY:
Inclusion Criteria

The inclusion criteria were patients of:

* more or equal to 18 years of age;
* Who have the virus with or without any co-morbidities;
* And who give consent to participate.

Exclusion Criteria:

* Patients who are imprisoned;
* And/or refuse to participate were excluded.

Disclaimer: prisoners were excluded as their confinement and lack of access will hinder them from receiving the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
KAP score (knowledge, attitude, and practices) | 6 months
  improving the overall nutrition-related knowledge and its reflection on patients' dietary knowledge, attitudes, and practices.
  The data was collected face-to-face using a questionnaire adapted from the relevant literature including questions related to nutrition knowledge, attitude, and practices (KAP) of HIV patients attending an outpatient clinic in India. This questionnaire assessed all 3 aspects, where the score ranges of knowledge, attitude, and practices are 0-14, 14-42, and 0-13, respectively. The total score of all three subsections ranges between 13-69 where a score between 13 and 32 represents poor KAP values, 33-51 average, and 52-69 good values. The original scores were modified in our study based on face and content validity results.
Improve in intake of immune boosting nutrients | 6 months
  Improving the food intake of immune-boosting foods and food groups (e.g.: fruits and vegetables, protein-containing food groups).
  Two-non-consecutive days 24-hour dietary recalls was used both pre- and post-intervention to measure the intake of total calories and protein as well as nutrients of immune-boosting properties (Vitamin A, Vitamin C, Vitamin E, Vitamin D, Selenium, Zinc, omega 3 omega 6 fatty acids, Iron). Additionally, a qualitative food frequency questionnaire was developed from the literature on the immune-boosting food groups. It was used to measure the change in intake of the immune-boosting food groups pre- and post-intervention period. It covered 10 components (fruits, vegetables, animal-derived protein food sources, plant-based protein food sources, whole grains, nuts, seeds, probiotic-rich foods, herbs, plant-based monounsaturated fatty acids rich oils, plant-based polyunsaturated fatty acids rich oils).

SECONDARY OUTCOMES:
Improve in physical activity | in 6 months
  Improving the physical activity levels and anthropometric measurements of PLHIV.
  Physical activity level (active versus inactive) was determined using a questionnaire developed by the American College of Sports Medicine for assessing the physical activity level of patients in clinical settings, namely the "Physical Vital Sign Questionnaire". The physically active versus inactive status is determined following the Physical Activity Guidelines for Americans, 2023, which recommend a physical activity level for adults of 150 minutes of moderate-intensity physical activity and 2 days of muscle-strengthening activity.
  Any participant performing any kind of physical activity for 150 minutes/week as well as 2-3 days of muscle strengthening workouts is considered physically active. Any participant below 150 minutes/week and no strength training whatsoever is considered physically inactive.
Body mass index (BMI) reduction | 6 months
  The measurements of weight is kilograms and the height in centimeter will be aggregated to arrive at one reported value which is BMI in Kg/m^2.
Improving nutrition-related biochemical data | in 6 months
  Improving the nutrition-related biochemical lab values in relation to adjustment of patients' dietary and lifestyle factors.
  Biochemical measurements were collected from the patient's medical files pre- and post-intervention for both control and intervention group.
  Reference Range for each biochemical parameter:
  Viral load: Ref not detected (Negative) copies/mL. CD4: Ref 219 - 1,621 CELL/uL. Hemoglobin: Ref males 13.0 - 17.0 g/dL versus females 12.0-15.0 g/dL. ALT: Ref males 0-41 U/L versus females 0-31 U/L. AST: Ref males 0-40 U/L versus females 0-32 U/L. Creatinine: Ref: males 0.7-1.2 mg/dL versus females 0.5-0.9 mg/dL. Urea: Ref 12-40 mg/dL. HbA1c: Ref more than5.7% - 5.7-6.4% prediabetes - >=6.5 diabetes. eGFR: Ref more than 60 mL/min/1.73(2) VitaminD3: Ref 30-100 ng/mL. LDL: Ref less than 115 mg/dL HDL: Ref above40 mg/dL men, above 48 mg/dL women. Triglyceride: Ref less than 90 mg/dL

OTHER OUTCOMES:
Change of mental health through hospital anxiety and depression scale (HADS) | in 6 months
  Change of the overall mental health status of PLHIV.
  Screening of mental health was done using the questionnaire Hospital Anxiety and Depression Scale (HADS) used to assess the prevalence of anxiety and depression. A score of 0-7 is normal, 8-10 mild anxiety/depression, 11-14 moderate anxiety/depression, 15-21 severe anxiety/depression. A validated Arabic version of the questionnaire was used on Arabic-speaking patients. A HADS score on each sub-section above 11 is elevated and needs further assessment by a psychologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Health - Rashid Hospital, Dubai, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No